CLINICAL TRIAL: NCT00739648
Title: Phase 2, Randomized, Double-Blind, Placebo-Controlled, Study to Evaluate the Safety, Tolerability and Efficacy of MP-376 Inhalation Solution Administered for 5 Days Every 28 Days to Prevent Acute Exacerbations in High Risk COPD Patients
Brief Title: A Phase 2 Study of MP-376 to Prevent Acute Exacerbations in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Mpex-302
Record Dates: First submitted 2008-08-20; First posted 2008-08-22 (Estimated); Results first posted 2012-03-02 (Estimated); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Patients
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo inhaled twice daily via the PARI eFlow nebulizer for 5 consecutive days within a 28-day treatment cycle for up to 12 cycles
  Interventions: Drug: Placebo
- MP-376 240 mg Twice Daily (BID) (Experimental): MP-376 240 mg BID inhaled via the PARI eFlow nebulizer for 5 consecutive days within a 28-day treatment cycle for up to 12 cycles
  Interventions: Drug: MP-376

INTERVENTIONS:
Drug: MP-376 — MP-376 administered via inhalation for 5 consecutive days within 28-day treatment cycles for up to 12 cycles
  Other Names: Levofloxacin inhalation solution; Aeroquin
  Arms: MP-376 240 mg Twice Daily (BID)
Drug: Placebo — same frequency as study drug using the same method of delivery
  Other Names: MP-376 color-matched placebo
  Arms: Placebo

SUMMARY:
Patients with Chronic Obstructive Pulmonary Disease (COPD) suffer from frequent and recurrent acute exacerbations (AECB) which are associated with enormous healthcare expenditures and significant morbidity, specifically an increased risk of death, a decline in pulmonary function and a significant change in quality of life. Bacteria appear to have an important role in acute exacerbations in chronic bronchitis and COPD. Studies of acute exacerbations in COPD have shown a reduction in bacterial load with prolonged exacerbation-free interval. In addition, recent studies indicate that acquisition of a new strain of H. influenzae, M. catarrhalis, S. pneumoniae or P. aeruginosa are responsible for many of these exacerbations. Chronic inflammation and bacterial infection predispose many patients to frequent and recurrent acute exacerbations.

Mpex believes that intermittent administration of inhaled MP-376 in high risk patients will decrease the incidence of acute exacerbations by both by lowering the organism burden, and resultant inflammation, as well as pre-emptive eradication of any newly acquired bacterial strains.

DETAILED DESCRIPTION:
This study will be a Phase 2, multi-center, randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, and efficacy of MP-376 inhalation solution given daily for 5 days in a 28 day treatment cycle to COPD patients.

Study with completed results acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria (selected):

* > 40 years of age
* History of COPD
* Forced expiratory volume in 1 second (FEV1) </= 70% of predicted and FEV1/Forced vital capacity (FVC) </= 0.7 value at screening
* Have at least two acute exacerbation episodes in the proceeding year
* Clinically stable with no changes in health status within the last 30 days
* Lifetime smoking history of at least 10 pack-years
* Willing and able to use a daily electronic diary

Exclusion Criteria (selected):

* Use of any systemic or inhaled antibiotics within 30 days prior to baseline
* History of hypersensitivity to fluoroquinolones or intolerance with aerosol medication
* Creatinine clearance < 40 mg/ml/min, AST, ALT >/= 5 x upper limit of normal (ULN) or total bilirubin >/= 3 x ULN at Screening

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2008-10; Primary Completion 2010-01 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (39):
- United States (39):
  - Haleyville, Alabama
  - Hueytown, Alabama
  - Mobile, Alabama
  - Montgomery, Alabama
  - Glendale, Arizona
  - Phoenix, Arizona
  - Chula Vista, California
  - Lomita, California
  - Long Beach, California
  - Mission Viejo, California
  - Oceanside, California
  - Palo Alto, California
  - Riverside, California
  - San Diego, California
  - San Jose, California
  - Wheat Ridge, Colorado
  - Clearwater, Florida
  - DeBary, Florida
  - DeLand, Florida
  - Orlando, Florida
  - Savannah, Georgia
  - New Orleans, Louisiana
  - Taylor, Michigan
  - Omaha, Nebraska
  - Buffalo, New York
  - Ithaca, New York
  - Greenville, North Carolina
  - Columbus, Ohio
  - Maumee, Ohio
  - Toledo, Ohio
  - Medford, Oregon
  - Johnston, Rhode Island
  - Easley, South Carolina
  - Gaffney, South Carolina
  - Spartanburg, South Carolina
  - Union, South Carolina
  - San Antonio, Texas
  - Richmond, Virginia
  - Salem, Virginia

REFERENCES:
- [Derived] Leidy NK, Murray LT, Monz BU, Nelsen L, Goldman M, Jones PW, Dansie EJ, Sethi S. Measuring respiratory symptoms of COPD: performance of the EXACT- Respiratory Symptoms Tool (E-RS) in three clinical trials. Respir Res. 2014 Oct 7;15(1):124. doi: 10.1186/s12931-014-0124-z. PMID 25287629
- [Derived] Leidy NK, Murray LT, Jones P, Sethi S. Performance of the EXAcerbations of chronic pulmonary disease tool patient-reported outcome measure in three clinical trials of chronic obstructive pulmonary disease. Ann Am Thorac Soc. 2014 Mar;11(3):316-25. doi: 10.1513/AnnalsATS.201309-305OC. PMID 24432712

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo inhaled twice daily via the eFlow nebulizer for 5 consecutive days within a 28-day treatment cycle for up to 12 cycles
- MP-376 240 mg BID: MP-376 240 mg inhaled twice daily via the PARI eFlow nebulizer for 5 consecutive days within a 28-day treatment cycle for up to 12 cycles
Period: Overall Study
Arm/Group | Placebo | MP-376 240 mg BID
Started | 108 | 214
Completed | 82 | 161
Not Completed | 26 | 53
Not completed — Adverse Event | 3 | 15
Not completed — Withdrawal by Subject | 13 | 25
Not completed — Lost to Follow-up | 4 | 7
Not completed — Death | 2 | 0
Not completed — Do not know | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MP-376 240 mg BID | Total
Number analyzed (Participants) | 108 | 214 | 322
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (9.06) | 64.0 (9.14) | 63.8 (9.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 101 | 153
  Male | 56 | 113 | 169

OUTCOME MEASURES:

1. Primary Outcome: Exacerbation Rate
Description: The number of acute exacerbations per patient-year of study participation, where an acute exacerbation was defined as a deterioration in respiratory symptoms that required treatment with antibiotics, corticosteroids, hospitalization or a combination of those treatments.
Time Frame: From randomization to the patients final study visit (up to 12 months)
Population: modified intent to treat (MITT; patients who received at least one dose of study drug)
Measure: Mean (Standard Error); unit: exacerbation per patient year
Groups:
- Placebo: Placebo inhaled twice daily (BID) via PARI eFlow nebulizer for 5 consecutive days in each 28-day treatment cycle for up to 12 cycles
- MP-376 240 mg BID: MP-376 240 mg inhaled twice daily (BID)via PARI eFlow nebulizer for 5 consecutive days in each 28-day treatment cycle for up to 12 cycles
Arm/Group | Placebo | MP-376 240 mg BID
Number analyzed (Participants) | 108 | 214
exacerbation per patient year | 1.20 (0.15) | 1.31 (0.11)
Statistical Analysis 1: Comparison: Placebo vs MP-376 240 mg BID; Test type: Superiority or Other; p = 0.7282, Regression, Linear; negative binomial regression model; Odds Ratio (OR) = 1.09, 90% CI 2-sided [0.86 to 1.39]

2. Secondary Outcome: Duration of Acute Exacerbation
Description: From the beginning of antibiotics and/or systemic corticosteroids to the end of antibiotics and/or systemic corticosteroids, whichever was longer, for treatment of the first acute exacerbation
Time Frame: from randomization to the patient's final study visit (up to 12 months)
Population: MITT
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Placebo: Placebo inhaled BID via nebulization for 5 consecutive days within a 28-day treatment cycle for up to 12 cycles
- MP-376 240 mg BID: MP-376 240 mg inhaled BID via nebulization for 5 consecutive days within a 28-day treatment cycle for up to 12 cycles
Arm/Group | Placebo | MP-376 240 mg BID
Number analyzed (Participants) | 108 | 214
Days | 12.9 (12.11) | 11.6 (7.98)

3. Secondary Outcome: Percent Change in Forced Vital Capacity (FVC)
Description: The percent change in the amount of air a patient can inhale
Time Frame: from baseline to the conclusion of the fourth 28-day treatment cycle (4 months)
Population: MITT
Measure: Least Squares Mean (Standard Error); unit: Percent
Groups:
- Placebo: Placebo inhaled BID via nebulization for 5 consecutive days in a 28-day cycle for up to 12 cycles
- MP-376 240 mg BID: MP-376 240 mg inhaled BID via nebulization for 5 consecutive days in a 28-day cycle for up to 12 cycles
Arm/Group | Placebo | MP-376 240 mg BID
Number analyzed (Participants) | 108 | 214
Percent | 14.46 (6.18) | -0.77 (4.43)
Statistical Analysis 1: Comparison: Placebo vs MP-376 240 mg BID; Test type: Superiority or Other; p = 0.9768, Mixed Models Analysis; Median Difference (Final Values) = -15.2, 90% CI 2-sided [-27.8 to -2.66]

4. Secondary Outcome: Percent Change in Forced Expiratory Volume in 1 Second (FEV1)
Description: The percent change in the amount of air a patient can exhale in 1 second
Time Frame: from baseline to the conclusion of the fourth 28-day treatment cycle (4 months)
Population: MITT
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Placebo | MP-376 240 mg BID
Number analyzed (Participants) | 108 | 214
Percent | 14.76 (6.21) | 2.42 (4.45)
Statistical Analysis 1: Comparison: Placebo vs MP-376 240 mg BID; Test type: Superiority or Other; p = 0.9464, Mixed Models Analysis; Mean Difference (Final Values) = -12.3, 90% CI 2-sided [-24.9 to 0.26]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Placebo | MP-376 240 mg BID
Serious Adverse Events (participants affected / at risk) | 32/108 | 72/214
Other Adverse Events (participants affected / at risk) | 94/108 | 197/214
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=108) | MP-376 240 mg BID (N=214)
Condition Aggravated (General disorders) | 22 (31) | 39 (53) — Pulmonary exacerbation
Chest pain (General disorders) | 3 (4) | 4 (4)
Catheter site hematoma (General disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Edema (General disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 10 (10)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 2 (2)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Bursitis infective staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis C (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0)
Nocardiosis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aoritic stenosis (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Malignant hypertension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (2) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gsatrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 0 (0) | 1 (1)
Paresis (Nervous system disorders) | 1 (1) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (2)
Mental status change (Psychiatric disorders) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedureal hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cholecystitits (Hepatobiliary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=108) | MP-376 240 mg BID (N=214)
Condition aggravated (General disorders) | 58 (120) | 114 (247) — Pulmonary exacerbation
Edema peripheral (General disorders) | 7 (8) | 16 (16)
Chest pain (General disorders) | 6 (7) | 13 (14)
Chest discomfort (General disorders) | 6 (6) | 11 (11)
Sinusititis (Infections and infestations) | 13 (13) | 11 (13)
Pneumonia (Infections and infestations) | 5 (6) | 17 (24)
Urinary tract infection (Infections and infestations) | 8 (10) | 10 (11)
Dyspenea (Respiratory, thoracic and mediastinal disorders) | 18 (21) | 29 (42)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (16) | 24 (25)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 9 (9)
Pharynlaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 8 (8)
Dysgeusia (Nervous system disorders) | 3 (3) | 62 (91) — Taste complaint
Headache (Nervous system disorders) | 11 (11) | 16 (18)
Nausea (Gastrointestinal disorders) | 13 (113) | 24 (28)
Diarrhea (Gastrointestinal disorders) | 7 (7) | 13 (14)
Vomiting (Gastrointestinal disorders) | 3 (3) | 11 (12)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4) | 12 (18)
Insomnia (Psychiatric disorders) | 6 (6) | 14 (15)
Anxiety (Psychiatric disorders) | 6 (6) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No